CLINICAL TRIAL: NCT06154915
Title: Characterise the Immunological Response of Diabetic Patients With Chronic Foot Ulcers
Brief Title: Immune Cells in Diabetic Chronic Foot Ulcers
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Cecilia Morgantini, MD, PhD, Karolinska Institutet
Other Study IDs: 2022-01416
Record Dates: First submitted 2023-11-17; First posted 2023-12-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot; Immune Defect
MeSH Terms: conditions — Diabetic Foot | interventions — Undertreatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and foot ulcer biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healing Ulcer: The patients will be recruited from the doctors and the nurses of the foot clinic of Department of Endocrinology. A complete medical history and physical parameters will be collected, moreover a peripheral circulation status will assess at the time of the enrolment. During the first visit blood samples and a biopsy from the site of foot ulcers will be taken together with a picture of the ulcer. All patients will follow the medical treatments, as recommended by the multidisciplinary clinical team (for example revascularization or ulcer debriding). Intervals between visits will range between 4 to 8 weeks according to the usual medical routine. During visits 1, 2 and 3 the ulcers status will be documented by pictures, physical parameter collected, biopsies, ulcer fluid and blood samples will be taken for further analysis.
  At visit 3 the ulcers will be classified as "healing" if completely resolved or dramatically reduced (more than 50%), otherwise will be classified as "non-healing".
  Interventions: Other: medical treatments
- Non-Healing Ulcer: The patients will be recruited from the doctors and the nurses of the foot clinic of Department of Endocrinology. A complete medical history and physical parameters will be collected, moreover a peripheral circulation status will assess at the time of the enrolment. During the first visit blood samples and a biopsy from the site of foot ulcers will be taken together with a picture of the ulcer. All patients will follow the medical treatments, as recommended by the multidisciplinary clinical team (for example revascularization or ulcer debriding). Intervals between visits will range between 4 to 8 weeks according to the usual medical routine. During visits 1, 2 and 3 the ulcers status will be documented by pictures, physical parameter collected, biopsies, ulcer fluid and blood samples will be taken for further analysis.
  At visit 3 the ulcers will be classified as "non-healing" if not resolved or not dramatically reduced (more than 50%).
  Interventions: Other: medical treatments

INTERVENTIONS:
Other: medical treatments — All patients will follow the medical treatments, as recommended by the multidisciplinary clinical team (for example revascularization or ulcer debriding) according to the best standard of care

SUMMARY:
The goal of this observational study is to learn about the role of immune cells in patients with diabetes and chronic foot ulcers. Researchers will compare blood and tissue samples of patients with diabetes and a foot ulcer that is healing or healed compared to those diabetic patients where the foot ulcers is not healing (chronic ulcer).

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) requires frequent hospital visits, anti-biotic therapies, and surgical procedures. Not only this approach has debilitating consequences for patients and enormous costs for the health care system, but it is often not sufficient to prevent lower limb amputation. The immunological response in wound healing is mainly orchestrated by recruited monocytes and skin macrophages. The current hypothesis is that hyperglycaemia sustains an activated macrophages' phenotype that inhibits wound healing. However, well controlled diabetes is not associated with better healing, and not all the diabetic patients develop chronic foot ulcers. In this project, the investigators aim to characterize the immunological response of patients with DFU to discover new therapeutic targets for the treatment of chronic wounds. The investigator suggest that an altered metabolic local environment can re-program monocytes/macrophages towards dysfunctional phenotypes unable to accomplish the healing process. Here, by using a longitudinal study cohort combined with clinical information, transcriptomic and proteomic analysis at single cell level, researchers will characterize the landscape of monocytes/macrophage populations involved in healing, and non-healing, foot ulcers. Functional validation will be performed in human skin organoids. My group's unique access to patient material combined with cutting-edge methodologies provides an exceptional platform to identify genes and pathways involved in chronic DFU.

ELIGIBILITY:
Inclusion Criteria:

* diabetes with diabetic foot ulcer

Exclusion Criteria:

* impaired cognitive function
* on-going immune suppressive treatment
* diagnosed active cancer
* cancer treatment
* known chronic inflammatory disease

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with one or more foot ulcer.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the longitudinal signature of circulating monocytes in the healing process of diabetic patients | 4 years
  An aliquot of peripheral blood mononuclear cells obtained from patients at the first visit will be used to perform single-cell RNA-sequencing. Transcriptomic results of patients with healing ulcers will be compared with those with non-healing ulcers in order to identify different circulating monocytes populations only present in non-healing diabetic patients.
Determine the functional contribution of macrophages to diabetic chronic foot ulcers | 4 years
  A freshly taken punch biopsy take from patient at visit 1 will be dissociated to a cell suspension. Single cell RNA sequencing analysis will be performed on these cells in order to study different cell populations. Bioinformatic analysis of sequenced data will identify macrophage's population, map cell heterogeneity and identify specific cell signature of healing compared to non-healing ulcers.
  Moreover, by comparing the transcriptomic signature of the cell populations in the tissue with circulating monocytes population defined in aim 1, researchers will verify whether specific populations are already present in circulation or appearing once the cells are in the tissue, or derived skin-resident macrophages.

CONTACTS AND LOCATIONS:
Overall Officials: cecilia Morgantini, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual participants data completely anonymised regarding trascriptomic and proteomic results will be shared in public repository